CLINICAL TRIAL: NCT03050021
Title: Risk Factors for Delirium in Critically Ill Surgical Patients
Status: Completed | Type: Observational
Sponsor: Suk-Kyung (Other)
Responsible Party: Sponsor-Investigator, Suk-Kyung, Associate Professor in General Surgery, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: 2014-0251
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Delirium; Intensive Care Unit Syndrome
Keywords: Delirium; Intensive care unit
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium positive: delirium patients in critically ill surgical patients
- Delirium negative: non delirium patients in critically ill surgical patients

SUMMARY:
Delirium is characterized by changes in mental status, inattension, disorganized thinking, and altered consciousness. Prevalence of delirium in critically ill patients has varied from 20~80% depending on the severity of illness. Despite its high prevalence, delirium is often under-recognized by clinicians due to the difficulties in diagnosis and no interest. Delirium is associated with increased mechanical ventilation days, hospital length of stay, and mortality. The purpose of this study is to analyze the prevalence of delirium and risk factors for delirium in critically ill surgical patients.

DETAILED DESCRIPTION:
The investigators performed a prospective cohort study involving the patients admitted to surgical ICU between april 2013 and august 2013.

The included patients were assessed independently by trained ICU nurses using the confusion Assessment Method for the ICU (CAM-ICU). The patients were recorded general characteristics, disease-related factors, and treatment and environment-related factors. Data were analyzed by SPSS 12.0 software, using t-test, Fisher's exact test and logistic regression.

ELIGIBILITY:
Inclusion Criteria:

1. Above RASS -3 paitent
2. Verbally or nonverbally communication possible patients

Exclusion Criteria:

1. Under age 18
2. Neurological disorder e.g.) Brain injury, dementia and traumatic brain injury
3. Readmitted to ICU
4. History of delirium
5. Transplanted; isolation is required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted to the surgical ICU from April to August 2013 and had the ability to express themselves verbally or nonverbally.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2013-08-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Prevelance of delirium | with in 6month in SICU
  Analyses were performed to delirium prevelance of SICU Patients

SECONDARY OUTCOMES:
Risk factors associated with delirium | with in 6month in SICU
  Analyses were performed to compare patient, disease, treatment and environment-related factors

CONTACTS AND LOCATIONS:
Overall Officials: Suk-kyung Hong, Ph.D, Principal Investigator — University of Ulsan College of Medicine. Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Result] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Result] Pisani MA, Araujo KL, Van Ness PH, Zhang Y, Ely EW, Inouye SK. A research algorithm to improve detection of delirium in the intensive care unit. Crit Care. 2006;10(4):R121. doi: 10.1186/cc5027. PMID 16919169
- [Result] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Result] Hsieh SJ, Ely EW, Gong MN. Can intensive care unit delirium be prevented and reduced? Lessons learned and future directions. Ann Am Thorac Soc. 2013 Dec;10(6):648-56. doi: 10.1513/AnnalsATS.201307-232FR. PMID 24364769
- [Result] Rapp CG, Mentes JC, Titler MG. Acute confusion/delirium protocol. J Gerontol Nurs. 2001 Apr;27(4):21-33; quiz 62-3. doi: 10.3928/0098-9134-20010401-07. PMID 11915153
- [Result] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Result] Hunt JM. The cardiac surgical patient's expectations and experiences of nursing care in the intensive care unit. Aust Crit Care. 1999 Jun;12(2):47-53. doi: 10.1016/s1036-7314(99)70535-7. PMID 10624186
- [Result] Peterson JF, Pun BT, Dittus RS, Thomason JW, Jackson JC, Shintani AK, Ely EW. Delirium and its motoric subtypes: a study of 614 critically ill patients. J Am Geriatr Soc. 2006 Mar;54(3):479-84. doi: 10.1111/j.1532-5415.2005.00621.x. PMID 16551316
- [Result] Irish JT. Deciphering the physician-older patient interaction. Int J Psychiatry Med. 1997;27(3):251-67. doi: 10.2190/CQ97-Y82H-6P2E-9BJ4. PMID 9565727
- [Result] Gustafson Y, Berggren D, Brannstrom B, Bucht G, Norberg A, Hansson LI, Winblad B. Acute confusional states in elderly patients treated for femoral neck fracture. J Am Geriatr Soc. 1988 Jun;36(6):525-30. doi: 10.1111/j.1532-5415.1988.tb04023.x. PMID 2897391
- [Result] Micek ST, Anand NJ, Laible BR, Shannon WD, Kollef MH. Delirium as detected by the CAM-ICU predicts restraint use among mechanically ventilated medical patients. Crit Care Med. 2005 Jun;33(6):1260-5. doi: 10.1097/01.ccm.0000164540.58515.bf. PMID 15942341
- [Result] Kamdar BB, Needham DM, Collop NA. Sleep deprivation in critical illness: its role in physical and psychological recovery. J Intensive Care Med. 2012 Mar-Apr;27(2):97-111. doi: 10.1177/0885066610394322. Epub 2011 Jan 10. PMID 21220271
- [Result] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Result] Bross MH, Tatum NO. Delirium in the elderly patient. Am Fam Physician. 1994 Nov 1;50(6):1325-32. PMID 7942430